CLINICAL TRIAL: NCT01414920
Title: A Phase 2, Randomized, Placebo-Controlled, Factorial, Double-Blind, Double-Dummy, Parallel-Group, Multicenter Study to Determine the Efficacy and Safety of 25 mg and 50 mg of TAK-875 in Combination With Sitagliptin 100 mg in Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of TAK-875 in Combination With Sitagliptin in Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-875_202; U1111-1115-5044 (Registry Identifier: WHO)
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — TAK-875; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- TAK-875 25 mg QD (Experimental)
  Interventions: Drug: TAK-875
- TAK-875 50 mg QD (Experimental)
  Interventions: Drug: TAK-875
- Sitagliptin 100 mg QD (Experimental)
  Interventions: Drug: Sitagliptin
- TAK-875 25 mg QD + Sitagliptin 100 mg QD (Experimental)
  Interventions: Drug: TAK-875 and Sitagliptin
- TAK-875 50 mg QD + Sitagliptin 100 mg QD (Experimental)
  Interventions: Drug: TAK-875 and Sitagliptin

INTERVENTIONS:
Drug: Placebo — TAK-875 and sitagliptin placebo-matching tablets, orally, once daily for up to 12 weeks.
  Arms: Placebo QD
Drug: TAK-875 — TAK-875 25 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: TAK-875 25 mg QD
Drug: TAK-875 — TAK-875 50 mg, tablets, orally, once daily for up to 12 weeks.
  Arms: TAK-875 50 mg QD
Drug: Sitagliptin — Sitagliptin 100 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: Januvia
  Arms: Sitagliptin 100 mg QD
Drug: TAK-875 and Sitagliptin — TAK-875 25 mg, tablets, orally, once daily and sitagliptin 100 mg tablets, orally, once daily for up to 12 weeks.
  Other Names: Januvia
  Arms: TAK-875 25 mg QD + Sitagliptin 100 mg QD
Drug: TAK-875 and Sitagliptin — TAK-875 50 mg, tablets, orally, once daily and sitagliptin 100 mg tablets, orally, once daily for up to 12 weeks.
  Other Names: Januvia
  Arms: TAK-875 50 mg QD + Sitagliptin 100 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of TAK-875, once daily (QD), in combination with sitagliptin QD in participants with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
TAK-875 is being developed at Takeda Global Research and Development, Inc. as an adjunct to diet and exercise to improve glycemic control in patients with T2DM.

Sitagliptin is an inhibitor of dipeptidyl peptidase-4 (DPP-4) approved as an adjunct to diet and exercise to improve glycemic control in adults with T2DM.

This study will investigate the effects of the combination of TAK-875 with a DDP-4 inhibitor on glycosylated hemoglobin reduction.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. The participant has either:

   * A historical diagnosis of Type 2 Diabetes (T2DM) without the chronic use (defined as >7 days) of anti-diabetic therapy within 8 weeks prior to Screening, and with at least an 8-week documented history of a diet and exercise plan at Screening OR,
   * A historical diagnosis of T2DM and stable on at least 1500 mg per day (or maximum tolerated dose) of metformin as monotherapy for at least 8 weeks at Screening. Participants on a stable dose of metformin who enter the study will continue on the same dose of metformin throughout the duration of the study.
4. The participant is a man or woman and aged 18 to 80 years, inclusive.
5. The participant's body mass index (BMI) (kg/m2) at Screening is ≥23 and ≤45.
6. The participant has an glycosylated hemoglobin (HbA1c) level at Screening between 7.5% and 10.0%, inclusive, if on metformin and between 7.5% to 10.9%, inclusive, if treated with diet and exercise alone.
7. The participant has a fasting plasma glucose level <14.4 mmol/L (<260 mg/dL), at Screening.
8. The participant has a fasting C-peptide concentration ≥0.26 nmol/L (≥0.8 ng/mL) at Screening.
9. If the participant takes any chronic, non-excluded medications, the dose of these medications must have been stable (no change in dose or drug) for at least 4 weeks prior to Screening.
10. The participant is able and willing to monitor their glucose levels with a home glucose monitor and consistently record his or her own blood glucose concentrations according to the given instructions.
11. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after last dose.
12. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.
13. A female participant of childbearing potential must have a negative serum human chorionic gonadotropin (HCG) pregnancy test at Screening (Visit 1) and at Placebo Run-in (Visit 2). A negative urine HCG pregnancy test is also required at Randomization (Visit 3), prior to administration of the first dose of double-blind study medication.
14. The participant's compliance with single-blind study medication during the run-in phase is at least 80% and does not exceed 120% based on tablet counts performed by the study staff.

Exclusion Criteria:

1. The participant has received any investigational compound within 4 weeks prior to Screening.
2. The participant has been enrolled in a previous TAK-875 study.
3. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. The participant has a history of hypersensitivity or allergies to TAK-875 or sitagliptin, or their excipients.
5. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 2 years prior to the Screening visit.
6. The participant has a history of cancer that has been in remission for <5 years prior to Screening (a history of basal cell carcinoma or stage 1 squamous cell carcinoma of the skin is allowed).
7. The participant has systolic blood pressure ≥150 mm Hg or diastolic pressure ≥90 mm Hg at Screening (Visit 1) or Baseline (Visit 3) (as confirmed by repeat measurement 30 minutes after initial measurement).
8. The participant has a creatine phosphokinase (CPK) level ≥5x the upper limit of normal (ULN) at Screening.
9. The participant has a hemoglobin level of ≤12 g/dL (120 gm/L) for men and ≤10 g/dL (100 gm/L) for women at Screening.
10. The participant has ALT and/or AST levels ≥2.5x ULN at Screening.
11. The participant has a total bilirubin level > ULN at Screening.
12. The participant has a serum triglyceride concentration ≥4.5 mmol/L (≥400 mg/dL) at Screening.
13. The participant has an estimated glomerular filtration rate ≤60mL/min using the Modification of Diet in Renal Disease (MDRD) equation at Screening.
14. The participant has a documented history or concurrent signs of uncontrolled (not euthyroid) thyroid disease (eg, autoimmune thyroid diseases such as Graves disease and Hashimoto thyroiditis or active thyroid nodules).
15. The participant has a history of pancreatitis.
16. The participant has a history of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
17. The participant has a history of gastric bypass surgery or has diabetic gastroparesis that in the investigator's opinion is moderate or severe and hence may impair absorption of study medication.
18. The participant has had coronary angioplasty, coronary stent placement, coronary bypass surgery, myocardial infarction, unstable angina pectoris, clinically significant abnormal electrocardiogram (ECG), cerebrovascular accident or transient ischemic attack within 6 months prior or at Screening.
19. The participant has a history of any hemoglobinopathy that may affect determination of HbA1c.
20. The participant has a positive test result for hepatitis B surface antigen and antibody to hepatitis C virus, and/or has known history of human immunodeficiency virus at Screening.
21. The participant has donated or received any blood products within 12 weeks prior to Screening.
22. The participant received medication prior to Screening as listed in the excluded Medications section.
23. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate an ova during such time period.
24. If male, the participant intends to donate sperm during the course of this study or for 30 days thereafter.
25. The participant has any other physical or psychiatric disease or condition that in the judgment of the investigator may affect life expectancy or may make it difficult to successfully manage and follow the participant according to the protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Glycosylated Hemoglobin (HbA1c) | Baseline and Week 12.
  The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 relative to baseline.

SECONDARY OUTCOMES:
Change from Baseline in Fasting Plasma Glucose | Baseline and Week 12.
  The change between the fasting plasma glucose value collected at week 12 relative to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director Clinical Science, Study Director — Takeda
Locations (80):
- United States (80):
  - Birmingham, Alabama
  - Brimingham, Alabama
  - Chandler, Arizona
  - Glendale, Arizona
  - Green Valley, Arizona
  - Mesa, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Buena Park, California
  - Irvine, California
  - Norwalk, California
  - Paramount, California
  - Rancho Cucamonga, California
  - San Ramon, California
  - Spring Valley, California
  - Vista, California
  - Walnut Creek, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Brandon, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Jupiter, Florida
  - Longwood, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Suwanee, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Valparaiso, Indiana
  - Crestview Hills, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Bangor, Maine
  - Elkridge, Maryland
  - Brockton, Massachusetts
  - Chelsea, Michigan
  - Kalamazoo, Michigan
  - Olive Branch, Mississippi
  - Berlin, New Jersey
  - Margate City, New Jersey
  - Toms River, New Jersey
  - Brooklyn, New York
  - Buffalo, New York
  - Calabash, North Carolina
  - Fuquay-Varina, North Carolina
  - Morehead City, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Lyndhurst, Ohio
  - Marion, Ohio
  - Willoughby Hills, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Broomall, Pennsylvania
  - Feasterville, Pennsylvania
  - Fleetwood, Pennsylvania
  - Cranston, Rhode Island
  - Chattanooga, Tennessee
  - Crossville, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - North Richland Hills, Texas
  - Pearland, Texas
  - San Antonio, Texas
  - Seattle, Washington